CLINICAL TRIAL: NCT06322420
Title: Mood-reactive Habitual Rumination and Changes During Behavioral Activation Treatment for Major Depression
Brief Title: Behavioral Activation for Depression and Habitual Rumination
Acronym: MoodHab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ragnar Pétur Ólafsson (Other)
Collaborators: The Icelandic Centre for Research (Unknown)
Responsible Party: Sponsor-Investigator, Ragnar Pétur Ólafsson, Professor at the Faculty of Psychology, University of Iceland, University of Iceland
Organization: University of Iceland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MoodHab
Record Dates: First submitted 2024-02-08; First posted 2024-03-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Active treatment provided to all participants in the study.
  Interventions: Behavioral: Behavioural Activation (BA)

INTERVENTIONS:
Behavioral: Behavioural Activation (BA) — Behavioural activation treatment delivered in this single arm study. Individual treatment given to all participants in 12 sessions over 11 weeks. All treatment components have been introduced by session 8 that defines minimum amount of treatment in the trial (i.e. 8 session completed).
  Behavioral Activation is a psychological treatment for depression focused on gradually re-engaging people with sources of reinforcement and reward in their environment by re-establish healthy patterns of activity, and replace avoidance behaviours with more adaptive behaviours.

SUMMARY:
Depressive rumination, a negative thinking style characterized by repetitive and passive thoughts about the causes, meanings, and consequences of one's feelings and distress, is often described as being a habitual response tendency that forms a vulnerability to depression. Behavioural Activation (BA) is an effective treatment for depression but little is known of mechanisms of changes during a successful treatment completion and for whom the treatment benefits the most. The main purpose of the study is to investigate whether habit-like mood-reactive rumination will change during Behavioral Activation treatment for current depression and mediates symptom changes in the treatment. Important moderators of change will also be investigated (i.e. history of early life stress and cognitive flexibility). We aim to provide individual BA treatment for up to 120 currently depressed participants (from 90 to 120 participants) in 12 treatment sessions over 11 weeks. Measures are obtained at pre-treatment, during treatment, at post-treatment and at 6 month follow up.

DETAILED DESCRIPTION:
Depressive rumination, a negative thinking style characterized by repetitive and passive thoughts about the causes, meanings, and consequences of one's feelings and distress, is often described as being a habitual response tendency that forms a vulnerability to depression. Behavioural Activation (BA) is an effective treatment for depression but little is known of mechanisms of changes during a successful treatment completion and for whom the treatment benefits the most. The main purpose of the study is to investigate whether habit-like mood-reactive rumination will change during Behavioral Activation treatment for current depression and mediates symptom changes in the treatment. Important moderators of change will also be investigated (i.e. history of early life stress and cognitive flexibility). We aim to provide individual BA treatment for up to 120 currently depressed participants (estimated number of participants is from 90 to 120) in 12 treatment sessions over 11 weeks. Measures are obtained at pre-treatment, during treatment (in sessions and during two assessment windows after session 4 and 8), at post-treatment and at 6 month follow up. Multimodal assessment of key constructs will be used in the study, including clinician ratings using semi-structured diagnostic interviews, self-report questionnaires, experimental tasks and ecological momentary assessment to capture moment-to-moment changes during the flow of daily life. Our main research questions are: 1) Does BA lead to reduction in depressive symptoms and diagnostic status, and are these symptom changes mediated by changes in habit-like mood-reactive ruminative thinking? 2) Are treatment gains and possible mediation of habit-like ruminative thinking, moderated by history of early-life stress and cognitive flexibility, that both have been established as predisposing factors for symptom onset in depression and are also know moderators of the development of rumination as a habit? 3) Does perceived control and reward-related responses increase during BA and are these changes associated with rumination as a habit? 4) Are gains during treatment maintained at 6-month follow up after treatment completion?

Moderators measured at pre-treatment: :

History of early life stess (total and physical/sexual/emotional abuse in particular), measured with the The Childhood Traumatic Event Scale (CTES) and The Adverse Childhood Experiences (ACEs) Questionnaire.

Cognitive flexibility: The Standard version of the Verbal Fluency Test (VFT), The Trail Making Test (TMT) and Digit-Span will be administered.

Mediators measured at pre-treatment, during treatment, post-treatment and follow up:

Depressive rumination will be measured with the brooding and reflective pondering subscales of the Ruminative Response Scale (RRS).

Habitual characteristics of ruminative thinking will be measured with the Habit Index of Negative Thinking (HINT).

Perceived control will be measured with the Pearlin Mastery Scale (PMS).

Reward-related responding will be measured with the Environmental Reward Observation Scale (EROS).

Level of activation will be measured with the Behavioral Activation for Depression Scale (BADS).

Selected items from the RRS, PMS, EROS and BADS are administered along the PHQ-9 at start of all treatment sessions in the study.

State ruminative thinking, perceived control, reward-related responding and level of activation will also be measured 8 times per day during ecological momentary assessment via smartphones for six days at pre-treatment and post-treatment and for three days at two assessment windows during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Current major depressive episode according to the DSM-5 diagnostic criteria evaluated with the DIAMOND diagnostic interview, that is considered to be the primary diagnosis.
2. Sore of 14 or higher on Becks Depression Inventory-II (BDI-II) that measures severity of symptoms of depression past 2 weeks.
3. Participants are between 18 and 65 years of age at start of study.
4. Satisfactory understanding of the Icelandic language to complete measures in the study.
5. Completion of pre-treatment assessment that includes 2 visits to researchers and a 6-day ecological momentary assessment.

Exclusion Criteria:

1. Current or past manic or hypomanic episodes according to the DSM-5 diagnostic criteria evaluated with the DIAMOND diagnostic interview.
2. Current or past psychotic disorders according to the DSM-5 diagnostic criteria evaluated with the DIAMOND diagnostic interview.
3. Presence of substance abuse within the last 12 months according to the DSM-5 diagnostic criteria evaluated with the DIAMOND diagnostic interview.
4. Presence of active and serious suicidal thoughts or a suicidal attempt in the previous 2 months.
5. Unstable medical treatment for depression (type of drug and/or dosing) during past two months at pre-treatment assessment.
6. Recent psychotherapy within the past month at pre-treatment assessment or active psychotherapy during study participation.
7. Cognitive impairments or severe physical illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Symptom severity measured by the BDI-2 | 2 weeks
  Severity of depressive symptoms as defined by BDI-2 (self-report rating). The BDI-2 will be administrated pre- and post treatment as a primary outcome measure.
  Additionally it will also be administrated after session 4 and session 8 and in a follow up measure 6 months after treatment ends.
  The BDI-2 is a 21 item self report scale. Each item is answered with a 4 point likert scale (0-3). The total score ranges from 0-63.
  Treatment response is defined as at least a 50% reduction in total symptom severity
Disorder severity assessed with the DIAMOND diagnostic interview - Major Depressive Disorder | 2 weeks
  The DIAMOND interview is intended to be used with adults (age 18 and up) with known or suspected Mood, Anxiety, or Obsessive- Compulsive and Related Disorders. The DIAMOND provides information on the diagnostic status and current severity for all disorders assessed in the interview according to DSM-5 criteria.
  This outcome is defined as severity (distress/impairment) of Major Depressive Disorder on a scale from 1-7 (normal, borderline, mild, moderate, marked, severe or extreme) at post-treatment (compared to pre-treatment assessment) assessed by an interviewer using the DIAMOND.
Diagnostic status assessed with the DIAMOND diagnostic interview - Major Depressive Episode | 2 weeks
  The DIAMOND interview is intended to be used with adults (age 18 and up) with known or suspected Mood, Anxiety, or Obsessive- Compulsive and Related Disorders. The DIAMOND provides information on the diagnostic status and current severity for all disorders assessed in the interview according to DSM-5 criteria.
  This outcome is defined as presence (or absence) of Major Depressive Episode in the past two weeks at post-treatment (compared to pre-treatment assessment), assessed by an interviewer using the DIAMOND.

SECONDARY OUTCOMES:
Symptom severity measured on the PHQ-9 | 1 week
  Severity of depressive symptoms measured with the PHQ-9 at post-treatment. The PHQ is as a 9 item self-administered measre for the assessment of the severity of depressive symptoms. Each item is answered with a 4 point likert scale (0-3). The total score ranges from 0-27.
  Treatment response is defined as at least a 50% reduction in total symptom severity.
Momentary negative and positive affectivity using items from the PANAS (Positive and Negative Affect Schedule) | 6 days
  Changes in momentary negative and positive affectivity using EMA (Ecological Momentary Assessment) via smartphones measured at post-treatment.
  Participants answer 8 multiple choice questions (1-5) eight times per day for six days (pre- and post treatment). Four items represent negative affectivity (NA) and four positive affectivity (PA). In the research group's previous studies, six of the items were used to calculate NA and PA scores, three for NA and three for PA. Consistent with previous research, three items will be used for each scale, thus total score for each scale can range from 3-15.
  Additionally the EMA measures will be administrated twice while treatment is ongoing, after session 4 and session 8, where the questions will be answered eight times per day for three days.
Diagnostic status assessed with the DIAMOND diagnostic interview at follow -up - Major Depressive Episode | 2 weeks
  The DIAMOND interview is intended to be used with adults (age 18 and up) with known or suspected Mood, Anxiety, or Obsessive- Compulsive and Related Disorders. The DIAMOND provides information on the diagnostic status and current severity for all disorders assessed in the interview according to DSM-5 criteria.
  This outcome is defined as presence (or absence) of Major Depressive Episode in the past two weeks at 6 months follow-up after end of treatment (compared to pre-treatment assessment), assessed by an interviewer using the DIAMOND.
Diagnostic status assessed with the DIAMOND diagnostic interview at follow-up- Major Depressive Disorder | 6 months
  The DIAMOND interview is intended to be used with adults (age 18 and up) with known or suspected Mood, Anxiety, or Obsessive- Compulsive and Related Disorders. The DIAMOND provides information on the diagnostic status and current severity for all disorders assessed in the interview according to DSM-5 criteria.
  This outcome is defined as presence (or absence) of Major Depressive Disorder in the past 6 months at 6 months follow-up after end of treatment.
The Quality of Life Scale (QOLS) | The QOL asks about how people experience their quality of life in the present, it will bee submitted through study completion, an average of 9 months, pre treatment, post treatment and in a 6 month follow up.
  The QOLS at post-treatment is a 16-item instrument that measured quality of life on a scale from 1-7 and the total score can range is from 16-112.

OTHER OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | 2 weeks
  The GAD-7 includes 7 items that assess symptoms of anxiety. Each item is answered on a four point likert scale from 0 to 3, total score range from 0-21. Measured at post-treatment and follow-up.
The Snaith-Hamilton Pleasure Scale (SHAPS) | 2 weeks
  The SHAPS measures anhedonia, the inability to experience pleasure and is a 14-item self-report questionnaire. Each question is on a scale from 0-3, total score range from 0-42. Measured at post-treatment and follow-up.
Beck Anxiety Inventory (BAI) | 1 week
  BAI is a self-report measure of severity of anxiety consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63. Measured at post-treatment and follow-up.
The Ruminative Response Scale (RRS) | The RRS asks about peoples rumination in the present, it will bee submitted through study completion, an average of 9 months, pre treatment, in treatment, post treatment and in a 6 month follow up.
  The RRS is be used to measure rumination tendencies. RRS includes 22 items that describe responses to depressed mood. These responses are self-focused, symptom-focused, and focused on the possible consequences and causes of their mood. Measured at post-treatment and follow-up.
The Pearlin Mastery Scale (PMS) | The PMS asks about how people regard their perceived control in the present, it will bee submitted through study completion, an average of 9 months, pre treatment, in treatment, post treatment and in a 6 month follow up.
  The PMS measures the extent to which an individual regards their life chances as being under their personal control rather than fatalistically ruled. It is a 7 item scale and the total score ranges from 7 to 35. Measured at post-treatment and follow-up.
The Environmental Reward Observation Scale (EROS) | 4 weeks
  The EROS contains 10 items that assess self-observed environmental reward that is essential for increasing response-contingent positive reinforcement. The total score range is 10-40. Measured at post-treatment and follow-up.
Behavioral Activation for Depression Scale (BADS) | 1 week
  The BADS measures when and how people become activated over the course of BA treatment using 25 item scale with a total score range from 0-150. Measured at post-treatment and follow-up.
Habit Index of Negative Thinking (HINT) | The HINT asks about habitual charectaristics in the present, it will bee submitted through study completion, an average of 9 months, pre treatment, in treatment, post treatment and in a 6 month follow up.
  Habitual characteristics of ruminative thinking will be measured with the Habit Index of Negative Thinking (HINT).
  The HINT is a 12 item self-report scale that measures the degree to which negative thoughts occur frequently, are initiated without awareness, are unintended, are difficult to control, and are self-descriptive in the present moment.
  The total score range is from 12-84. Measured at post-treatment and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ragnar P Ólafsson, PhD, Study Chair — University of Iceland
Locations (1):
- University of Iceland, Reykjavik, Iceland, Iceland

IPD SHARING:
Plan to Share IPD: Undecided